CLINICAL TRIAL: NCT05284552
Title: The Effect of Tinzaparin on Biomarkers in FIGO Stage III-IV Ovarian Cancer Patients Undergoing Neoadjuvant Chemotherapy - A Randomized Pilot Study
Brief Title: Tinzaparin And Biomarkers After Neoadjuvant Treatment of Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Region Jönköping County (Other Government); Västervik Hospital (Other); Vastra Gotaland Region (Other Government); Region Västerbotten (Other Government)
Responsible Party: Principal Investigator, Preben Kjolhede, MD, professor, Professor, senior consultant, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The TABANETOC-trial; 2021-000135-31 (EudraCT Number)
Record Dates: First submitted 2022-02-06; First posted 2022-03-17 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Tinzaparin; Neoadjuvant chemotherapy; FIGO stage III-IV
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Drug: Tinzaparin (Innohep®), solution for injection. Administration form: Subcutaneous injection. Dosage: 4500 IU (for subjects weighing below 90 kg) or 8000 IU (for subjects weighing 90 kg and above) daily for 21-28 weeks.
  Interventions: Drug: Tinzaparin Injectable Solution
- Control Arm (No Intervention)

INTERVENTIONS:
Drug: Tinzaparin Injectable Solution — Subcutaneous injection
  Other Names: Innohep®
  Arms: Intervention Arm

SUMMARY:
Background:

Previous findings have indicated antineoplastic properties of tinzaparin (Innohep®), a commonly used anti-coagulant. Earlier studies have mainly investigated the antineoplastic effects of tinzaparin in animal models and in human cell-lines. In this pilot study the aim is to examine the potential antitumoral effects of tinzaparin in vivo in women with epithelial ovarian cancer (EOC).

Study objectives:

Primary objective: The primary objective of the study is to evaluate the effects of tinzaparin on changes in levels of CA-125 in EOC patients who receive neoadjuvant chemotherapy (NACT).

Secondary objectives: The secondary objective of the study is to explore the impact of tinzaparin on the dynamic of a spectrum of immunological and coagulation factors in EOC patients who receive NACT. Besides, the compliance of tinzaparin injections and adverse events caused by tinzaparin will be described.

DETAILED DESCRIPTION:
This is an open randomized controlled clinical pilot trial (Phase II). The study includes women with the International Federation of Obstetrics and Gynecology (FIGO) stage III-IV EOC selected for neoadjuvant chemotherapy (NACT) and without signs of thromboembolic disease or ongoing treatment of thromboembolic disease. The women will be allocated 1:1 to treatment with tinzaparin 4500 IU/8000 IU (dose depending on woman's weight) subcutaneously once daily or no tinzaparin. The treatment group starts tinzaparin when the primary treatment (chemotherapy) starts. The control group will not receive tinzaparin or other low molecular weight heparin preparations. The NACT consists of carboplatin and paclitaxel, given according to the standard regimen with cycle repeats every 21 days. Pre-treatment, before every cycle of chemotherapy, before delayed primary debulking surgery (DPDS) and three weeks after the last cycle of chemotherapy venous blood samples will be taken for measuring the biomarkers hemoglobin, platelets, leucocytes, C-reactive protein (CRP), albumin, cancer antigen-125 (CA-125), Tissue Factor, D-dimer, soluble P-selectin, thrombin-antithrombin complex and thrombin generation potential. Furthermore, a panel of 92 inflammation-associated proteins will be analyzed by a by a high-sensitivity Proximity Extension Assay at baseline, visit 5 and visit 8 or 9. After three cycles of NACT, the patient will be evaluated clinically and with imaging diagnostics in order to determine whether the patient should undergo DPDS. In the investigators´ setting, > 80% of patients receiving NACT for EOC undergo DPDS. After DPDS, all patients will be treated with tinzaparin for 28 days according to clinical practice concerning postoperative thromboembolic prophylaxis and thereafter continue the chemotherapy for additional two-three courses. The participants who were allocated to tinzaparin during the NACT will continue the tinzaparin after ending the postoperative thromboembolic prophylactic tinzaparin treatment for additional 2-3 courses. The biomarkers will be measured preoperatively and four weeks postoperatively after DPDS and then before each course of chemotherapy given during the primary treatment. The women who do not undergo surgery will remain included in the study for the following three cycles of chemotherapy. Thus, the total study period constitutes 22-29 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written consent to participate in the study.
* Age 18 and above
* Epithelial ovarian, fallopian tube or peritoneal cancer, or abdominal cancer where a biopsy indicates an origin from the ovary, fallopian tube or peritoneum.
* Histology diagnosis of either high grade serous carcinoma, endometrioid carcinoma or clear cell carcinoma.
* FIGO stage III-IV disease.
* Selected for NACT with platinum double regimen at a multidisciplinary conference at Department of Oncology at Linköping University Hospital
* Receive treatment at either of the University Hospital in Linköping, or the hospitals in Jönköping (Ryhov Hospital), Eksjö (Highland Hospital, Eksjö), Västervik (Västervik hospital), Kalmar (County Hospital, Kalmar), Värnamo (Värnamo hospital).
* Planned for platinum doublet regimen.
* Prior to start of NACT pregnancy should be ruled out by menstrual history or in unclear cases by a urine human chorionic gonadotropin (hCG) test.
* Women of childbearing potential should use a safe birth control method (combined hormonal contraception, progesterone only hormonal contraception, intra uterine device, bilateral tubal occlusion, vasectomized partner, sexual abstinence, male or female condom, diaphragm with spermicide).
* World Health Organization (WHO) Performance Status 0-1
* Weight 50-150 kg
* CA-125-level ≥250 kIU/L at diagnosis

Exclusion Criteria:

* Concomitant treatment with heparins, low molecular weight heparins, warfarin or nonvitamin K antagonist oral anticoagulants. Platelet inhibitors are allowed.
* Treatment with heparins, low molecular weight heparins or non-vitamin K antagonist oral anticoagulants within the last year.
* Known or suspected allergies against any product included in the study
* Ongoing pregnancy, independent of gestational age. Breastfeeding or planned pregnancy
* EOC disclosed at Cesarean section
* Abdominal surgery or other major surgery within the last year
* Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of study participation
* Treatment or disease which, according to the investigator, can affect treatment or study results
* Known brain metastasis
* Participation or recent participation (within the last 30 days) in a clinical study with an investigational product
* Ongoing treatment of thromboembolic disease.
* Thromboembolic disease within the last year.
* Hypersensitivity to the active substance (tinzaparin) or any of the excipients.
* Serious hemorrhage or conditions predisposing to serious hemorrhage. Serious hemorrhage is defined as fulfilling any one of these three criteria:

  1. occurs in a critical area or organ (e.g. intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, intra-uterine or intramuscular with compartment syndrome),
  2. causes a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more, or
  3. leads to transfusion of two or more units of whole blood or red blood cells.
* Severe coagulation disorder.
* Acute gastro duodenal ulcer.
* Septic endocarditis.
* Previous heparin-induced thrombocytopenia.
* WHO Performance Status >1.
* Platinum single regimen
* Estimated glomerular filtration rate (E-GFR) <30ml/min (analyzed no more than 14 days before start of treatment with investigational product)
* Platelets <100 x10^9/L (analyzed no more than 14 days before start of treatment with investigational product)
* Treatment for other known malignancy within the last year (except basal cell carcinoma)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in serum levels of CA-125 | 14 weeks
  kIU/L

SECONDARY OUTCOMES:
Changes in serum levels of CA-125 | 21-28 weeks
  kIU/L
Changes in blood levels of hemoglobin | 21-28 weeks
  g/L
Changes in blood levels of platelets | 21-28 weeks
  x10^9/L
Changes in blood levels of leucocytes | 21-28 weeks
  x10^9/L
Changes in plasma levels of CRP | 21-28 weeks
  mg/L
Changes in plasma levels of albumin | 21-28 weeks
  g/L
Changes in plasma levels of interleukin 6 | 21-28 weeks
  ng/L
Changes in plasma levels of vascular endothelial growth factor | 21-28 weeks
  µg/L
Self reported compliance to tinzaparin injections | 22-29 weeks
  Percent
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 22-29 weeks
  Number
Proportion of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 22-29 weeks
  Proportion constitutes the relative number in the group in percent
Objectively confirmed venous thromboembolism (VTE), i.e. pulmonary embolism, lower-limb deep vein thrombosis or upper extremity deep vein thrombosis. Death due to VTE. | 22-29 weeks
  Number
Objectively confirmed venous thromboembolism (VTE), i.e. pulmonary embolism, lower-limb deep vein thrombosis or upper extremity deep vein thrombosis. Death due to VTE. | 22-29 weeks
  Percent

OTHER OUTCOMES:
Plasma levels of tissue factor | 21-28 weeks
  µg/L
Plasma levels of D-dimer | 21-28 weeks
  mg/L
Plasma levels of soluble P-selectin | 21-28 weeks
  µg/L
Plasma levels of thrombin-antithrombin complex | 21-28 weeks
  µg/L
Thrombin generation potential | 21-28 weeks
  lag time (min)
Thrombin generation potential | 21-28 weeks
  endogenous thrombin generation potential (nmolar*min)
Thrombin generation potential | 21-28 weeks
  peak nmol/L
Olink Target 96 Inflammation - plasma levels a panel of 92 inflammation associated proteins | 21-28 weeks
  All 92 inflammation associated proteins are measured in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Preben Kjölhede, MD, PhD, Study Chair — University Hospital, Linkoeping; Gabriel Lindahl, MD, PhD, Study Chair — University Hospital, Linkoeping; Anna-Clara Spetz Holm, MD, PhD, Study Chair — University Hospital, Linkoeping; Anna Karlsson, MD, Study Chair — University Hospital, Linkoeping
Locations (8):
- Sweden (8):
  - Department of Obstetrics and Gynecology, Highland Hospital, Eksjö
  - Department of Oncology, Sahlgrenska University Hospital, Gothenburg
  - Department of Obstetrics and Gynecology, Ryhov County Hospital, Jönköping
  - Department of Oncology, Linköping University Hospital, Linköping
  - Department of Obstetrics and Gynaecology, Norrland University Hospital, Umeå
  - Department of Obstetrics and Gynecology, Värnamo Hospital, Värnamo
  - Department of Obstetrics and Gynecology, Västervik Hospital, Västervik
  - Department of Obstetrics and Gynecology, University Hospital, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT05284552/Prot_SAP_000.pdf